CLINICAL TRIAL: NCT06108700
Title: Ergonomic Risk Assessment for Musculoskeletal Disorders in Office Workers Turkish Version, Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_08
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, there is a relationship between the increase in the use of electronic devices such as smartphones or tablets and musculoskeletal disorders. Different usage styles of various electronic devices such as laptops, smartphones and tablets affect the risk factors that may be related to musculoskeletal disorders in office workers. In addition to the use of electronic devices, the posture of the office worker's head, waist and hands while sitting are among the risk factors. Parameters such as the features of the chair he is sitting on, the height and distance of the table affect the person's posture. Evaluation of these factors is important in preventing musculoskeletal disorders.

The Ergonomic Risk Assessment for Musculoskeletal Disorders in Office Workers was developed by Kluay-On et al. in 2022 and its validity and reliability were established. The aim of our study is to culturally adapt the Ergonomic Risk Assessment for Musculoskeletal Disorders in Office Workers into Turkish and to examine its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Being an employee of Tokat Gaziosmanpaşa University
* Being an office worker

Exclusion Criteria:

* Not being an office worker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Office workers at Tokat Gaziosmanpaşa University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Ergonomics Risk Assessment for Musculoskeletal Disorders in Office Workers | Baseline
  Ergonomics Risk Assessment for Musculoskeletal Disorders in Office Workers consists of a total of 10 questions and 3 subsections. The first part includes 3 items related to health status, such as history of neck and low back pain and electronic device behaviors, which evaluate individual factors. In the second section, the physical factors section, there are 5 items related to working posture. In the last section, psychosocial factors, there are 2 items related to mental fatigue.
Ergonomics Risk Assessment for Musculoskeletal Disorders in Office Workers | After 1 week (retest)
  Ergonomics Risk Assessment for Musculoskeletal Disorders in Office Workers consists of a total of 10 questions and 3 subsections. The first part includes 3 items related to health status, such as history of neck and low back pain and electronic device behaviors, which evaluate individual factors. In the second section, the physical factors section, there are 5 items related to working posture. In the last section, psychosocial factors, there are 2 items related to mental fatigue.
New York Posture Rating Chart | Baseline
  In the evaluation, five (5) points are given if the person's posture is correct, three (3) points are given if the posture is moderately impaired, and one (1) point is given if the posture is seriously impaired. The total maximum score obtained as a result of the test is 65 and the minimum score is 13.
Short Form 36 | Baseline
  The subscales of the scale are: physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems 31 (3 items), mental health (5 items), energy (4 items). item), pain (2 items) and general perception of health (5 items). Subscales evaluate health between 0 and 100, with 0 indicating the lowest quality of life and 100 indicating the highest quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)